CLINICAL TRIAL: NCT06817876
Title: Connecting Caregivers With Community Services: The Care Buddy Platform
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Collaborators: Agency for Science, Technology and Research (A*STAR) (Other Government); Khoo Teck Puat Hospital (Other)
Responsible Party: Principal Investigator, Chetna Malhotra, Associate Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022-309
Record Dates: First submitted 2025-02-05; First posted 2025-02-10 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CareBuddy (Experimental): Caregivers of person with dementia who will be randomized in this arm will have access to the CareBuddy mobile app on their phone. They will be using this app for 1 year and will be followed up every 2 months.
  Interventions: Device: Care Buddy
- Usual care (No Intervention): Caregivers of person with dementia who will be randomized in this arm will continue usual care for their loved one. They will be enrolled for 1 year and will be followed up every 2 months.

INTERVENTIONS:
Device: Care Buddy — Care Buddy mobile intervention will be a one-stop solution for caregivers of dementia patients and help them in their care-giving journey by providing them solutions to manage behavioural problems, physical conditions of their loved one. The app will be multi-component and will provide tools for the caregiver to manage their stress and burden. It will provide information on dementia, list of service providers, information on grief, financial support. This app will provide a platform for all enrolled caregivers to chat with each other and provide social support.
  Arms: CareBuddy

SUMMARY:
The study aims to develop a mobile-app (Care Buddy) which will be a one-stop integrated source of information and technology-based solutions for caregivers of people with dementia (PWDs). Study aims to bring caregivers into closer partnerships with the wider ecosystem (e.g., healthcare practitioners, community services, peer support, and care service providers) which will ultimately improve outcomes for both PWDs and their caregivers.

DETAILED DESCRIPTION:
This is a 5-year study with various stages: 1) proof-of-concept stage to design and develop the Care buddy intervention, 2) proof-of-value stage to assess the feasibility, acceptability and satisfaction with the Care buddy intervention among informal caregivers of PWDs, 3) test-bedding stage to assess the efficacy and cost-effectiveness of the Care buddy intervention versus usual care among informal caregivers of PWDs with help of a multi-centre 2-arm RCT and 4) deployment stage to scale up the intervention at multiple centres across Singapore, monitor its adoption and outcomes and assess any organizational and individual barriers to adoption.

By the end of the proposed five-year project, investigators aim to develop and evaluate the technology as well as achieve widespread adoption among caregivers of PWDs. Investigators want to enable easy access to information, provide decisional and social support, improve the reach and uptake of existing community service providers, and assist with coordination among multiple informal and professional caregivers through the journey of dementia caregiving and into the bereavement phase.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for patients are

  1. Singaporean/Permanent residents
  2. Age 21 years of age or older
  3. Main person or one of the main persons involved in making decisions regarding treatment patient receives or responsible for ensuring the well-being of the patient
  4. An active primary caregiver for at least 6 months, and planning to remain the primary caregiver for the next 2 years
  5. Is a family member of the patient with dementia
  6. Can read and write in English
  7. Accessible by telephone to schedule interviews
  8. Has familiarity with use of technology (e.g., computers, tablets, or internet) and is able to complete surveys, forms using digital technology
  9. Intact cognition determined through the Abbreviated Mental Test (AMT) for those who are ≥ 65 years old.
  10. Caregivers who score >=9 on the 6-item Zarit Burden scale

Exclusion Criteria:

* Caregivers of patients staying in nursing home or other long-term care facility with no intention of being discharged will not be eligible however, if the patient is admitted to respite care for short/long term duration after being recruited, caregivers can continue to participate.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Caregiver Psychological well-being | 1 year from data collection
  Flourish - range - 8 - 56, high score represents a person with many psychological resources and strengths
Caregiver social scale | 1 year from data collection
  Friendship scale - The score range is 0-24. A high score represents social connectedness and a score of "0" complete social isolation
Caregiver Dementia Knowledge | 1 year from data collection
  The Dementia Knowledge Assessment Tool - range - 0-21. High score equals to higher knowledge of dementia.
Caregiver Impact | 1 year from data collection
  Revised Memory & Behavior Problem checklist - range - 0-96 Higher score indicates increased impact.
Caregiver Burden | 1 year from data collection
  Zarit Burden scale - range 0-88. 0 - 21 little or no burden, 21 - 40 mild to moderate burden, 41 - 60 moderate to severe burden, 61 - 88 severe burden >34 - clinically significant burden.
Caregiver Stress | 1 year from data collection
  Perceived Stress Scale: Scoring: PSS scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the four positively stated items (items 4, 5, 7, & 8) and then summing across all scale items.

OTHER OUTCOMES:
Health care costs | 1 year from data collection
  Health care costs, hospitalizations and emergency room visits for caregivers and PWDs will be obtained from patient billing data.

CONTACTS AND LOCATIONS:
Locations (1):
- Duke-NUS, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No